CLINICAL TRIAL: NCT05051592
Title: Role of Circulating Tumour DNA (ctDNA) Testing in Assessing for Alterations of Primary Anti-Epidermal Growth Factor Receptor (EGFR) Resistance in RAS/RAF Wild-type Metastatic Colorectal Cancer Patients
Brief Title: Role of Circulating Tumour DNA Testing in Assessing for Alterations of Primary Anti-EGFR Resistance in RAS/RAF Wild-type Metastatic Colorectal Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/00339
Record Dates: First submitted 2021-09-08; First posted 2021-09-21 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: ctDNA; anti_EGFR; RAS/RAF wild-type metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample collected from patient for this study, tumour or normal tissue removed or biopsied as part of patient's routine care and body fluids (e.g. fluid lining the lungs or effusion or fluid lining the abdomen or ascites) removed as part of patient's clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to explore the clinical utility of circulating tumour DNA (ctDNA) in assessing for alterations of anti-epidermal growth factor receptor (EGFR) primary resistance in RAS and BRAF wild-type metastatic colorectal cancer (CRC) patients treated with anti-EGFR monoclonal antibodies (cetuximab / panitumumab) in combination with fluorouracil (FU)-doublet chemotherapy.

DETAILED DESCRIPTION:
A single blood sample (20mL) will be collected after the patient has given informed consent. The blood sample will be collected within 4 weeks prior to the patient starting chemotherapy. Blood samples collected will be processed in accordance with the Guardant360 Clinical Blood Collection Kit instructions (Guardant Health, Inc.).

Patient outcomes with respect to response rate, progression-free survival, overall survival, toxicities and other co-morbid conditions will be ascertained by medical record review conducted by the study personnel. Prospective clinical data that will be collected include: patient demographics, tumor stage and pathological tumor characteristics at diagnosis, laboratory data at diagnosis and serial pre-specified time points, imaging outcomes, chemotherapy information, date of recurrence, and date and cause of death.

Although the data will be censored at the study end-points, the patient's medical record will be reviewed indefinitely to follow the health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stage IV colon or rectal cancer who are RAS/BRAF wild-type by routine tumor profiling and who are beginning standard-of-care treatment with fluorouracil-based doublet chemotherapy in combination with anti-EGFR monoclonal antibodies. Prior treatment with adjuvant therapy is allowed if completed more than 6 months prior to relapse of disease.

Exclusion Criteria:

* Pregnant women will be excluded from the study.
* Patient unable to give informed consent will be excluded from the study.
* Patients who have previously received chemotherapy in the metastatic setting.
* Patients who have previously received adjuvant chemotherapy less than 6 months prior to relapse of metastatic disease.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed RAS/BRAF wild-type mCRC who are beginning standard-of-care treatment with fluorouracil-based doublet chemotherapy in combination with anti-EGFR monoclonal antibodies will be recruited into the study. These are patients who are cared for at the National University Cancer Institute, Singapore (NCIS), and identified through the colorectal surgery, medical oncology and multidisciplinary CRC tumour board at NCIS.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Detection rate of alterations of anti-epidermal growth factor receptor primary resistance using Circulating tumour DNA | One timepoint, within 4 weeks prior to starting of anti-EGFR therapy
  ctDNA analysis will be carried out using Guardant360 platform to identify subgroup of patients who have primary resistance to anti-EGFR therapy.

SECONDARY OUTCOMES:
Response rate | 1 year 6 months
  Response rate to treatment received as per standard care.
Progression-free survival | 1 year 6 months
  The time from commencement of cancer treatment to disease progression or death from any cause.
Overall survival | 1 year 6 months
  The length of time from start of treatment to death.
Adverse reactions experience by patient | 1 year 6 months
  Toxicities in patients who have primary resistance to anti-EGFR therapy will be collected and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Ean Chee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Cutsem E, Cervantes A, Adam R, Sobrero A, Van Krieken JH, Aderka D, Aranda Aguilar E, Bardelli A, Benson A, Bodoky G, Ciardiello F, D'Hoore A, Diaz-Rubio E, Douillard JY, Ducreux M, Falcone A, Grothey A, Gruenberger T, Haustermans K, Heinemann V, Hoff P, Kohne CH, Labianca R, Laurent-Puig P, Ma B, Maughan T, Muro K, Normanno N, Osterlund P, Oyen WJ, Papamichael D, Pentheroudakis G, Pfeiffer P, Price TJ, Punt C, Ricke J, Roth A, Salazar R, Scheithauer W, Schmoll HJ, Tabernero J, Taieb J, Tejpar S, Wasan H, Yoshino T, Zaanan A, Arnold D. ESMO consensus guidelines for the management of patients with metastatic colorectal cancer. Ann Oncol. 2016 Aug;27(8):1386-422. doi: 10.1093/annonc/mdw235. Epub 2016 Jul 5. PMID 27380959
- [Background] Morano F, Corallo S, Lonardi S, Raimondi A, Cremolini C, Rimassa L, Murialdo R, Zaniboni A, Sartore-Bianchi A, Tomasello G, Racca P, Clavarezza M, Adamo V, Perrone F, Gloghini A, Tamborini E, Busico A, Martinetti A, Palermo F, Loupakis F, Milione M, Fuca G, Di Bartolomeo M, de Braud F, Pietrantonio F. Negative Hyperselection of Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer Who Received Panitumumab-Based Maintenance Therapy. J Clin Oncol. 2019 Nov 20;37(33):3099-3110. doi: 10.1200/JCO.19.01254. Epub 2019 Sep 20. PMID 31539295
- [Background] Vanderlaan PA, Yamaguchi N, Folch E, Boucher DH, Kent MS, Gangadharan SP, Majid A, Goldstein MA, Huberman MS, Kocher ON, Costa DB. Success and failure rates of tumor genotyping techniques in routine pathological samples with non-small-cell lung cancer. Lung Cancer. 2014 Apr;84(1):39-44. doi: 10.1016/j.lungcan.2014.01.013. Epub 2014 Jan 28. PMID 24513263
- [Background] Alix-Panabieres C, Pantel K. Clinical Applications of Circulating Tumor Cells and Circulating Tumor DNA as Liquid Biopsy. Cancer Discov. 2016 May;6(5):479-91. doi: 10.1158/2159-8290.CD-15-1483. Epub 2016 Mar 11. PMID 26969689
- [Background] Merker JD, Oxnard GR, Compton C, Diehn M, Hurley P, Lazar AJ, Lindeman N, Lockwood CM, Rai AJ, Schilsky RL, Tsimberidou AM, Vasalos P, Billman BL, Oliver TK, Bruinooge SS, Hayes DF, Turner NC. Circulating Tumor DNA Analysis in Patients With Cancer: American Society of Clinical Oncology and College of American Pathologists Joint Review. J Clin Oncol. 2018 Jun 1;36(16):1631-1641. doi: 10.1200/JCO.2017.76.8671. Epub 2018 Mar 5. PMID 29504847
- [Background] Krebs MG, Metcalf RL, Carter L, Brady G, Blackhall FH, Dive C. Molecular analysis of circulating tumour cells-biology and biomarkers. Nat Rev Clin Oncol. 2014 Mar;11(3):129-44. doi: 10.1038/nrclinonc.2013.253. Epub 2014 Jan 21. PMID 24445517
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720